CLINICAL TRIAL: NCT06223295
Title: Effectiveness of Focal Therapy in Men With Prostate Cancer
Acronym: ENFORCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Isala (Other); Amsterdam UMC, location VUmc (Other); St. Antionius Hospital (Unknown); Hifu kliniek (Unknown); Dutch National Health Care Institute (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Nederlandse Vereniging voor Radiotherapie en Oncologie (Unknown); Wetenschapscommissie interventieradiologie/Nederlandse vereniging voor interventieradiologie (Unknown); Inspire2live (Unknown); Prostaatkankerstichting (Unknown); Nederlandse Vereniging voor Urologie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-16261
Record Dates: First submitted 2023-09-07; First posted 2024-01-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: prostate neoplasm; focal therapy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal therapy (Active Comparator): Patients in this group will receive focal therapy, i.e. TULSA, IRE or Hifu.
  Interventions: Procedure: Focal therapy
- Usual care (Active Comparator): Patients in this group will receive usual care for prostate cancer, i.e. radical prostatectomy or radiotherapy
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Focal therapy — Focal therapy selectively treats a specific part of the prostate while preserving the rest of the gland in men with prostate cancer.
  Focal therapy with ultrasound ablation (HIFU/TULSA) or irreversible electroporation (IRE) followed by an intensive MRI follow-up scheme at 12, 24, 36, 48 and 60 months, prostate biopsy at 12 months (and also when indicated) and PSA monitoring
  Other Names: TULSA; IRE; Hifu
  Arms: Focal therapy
Procedure: Usual care — standard radical treatment; prostatectomy or radiotherapy with follow-up according international guidelines (PSA monitoring and imaging when indicated).
  Other Names: Radical prostatectomy; Radiotherapy
  Arms: Usual care

SUMMARY:
In the Netherlands, most men with prostate cancer (PCa) are treated with radical whole-gland treatment, i.e. prostatectomy or radiotherapy. The burden of complications such as incontinence and erectile dysfunction associated with radical treatment is considerable. A recent systematic review by our group has shown that focal therapy of PCa seems to reduce the burden of treatment side-effects in men with intermediate-risk disease, maintaining their quality of life without compromising oncological effectiveness. The costs of side effects that can be prevented are estimated at €5456 per patient, resulting in total expected cost savings of about €22 million per year in The Netherlands. Furthermore, exploration of the benefit-risk balance under patients showed that they are willing to sacrifice some survival for an improvement in quality of life (QoL).

Focal therapy comprises a modern alternative to selectively treat a specific part of the prostate while preserving the rest of the gland. There is, however, a lack of high-quality evidence, and numerous papers therefore recommend to perform a multicenter randomized controlled trial (RCT). The RCT should have long-term follow-up, predefined assessment of cancer-specific and health-related QoL outcome measures, and economic evaluations to inform policymakers regarding cost-effectiveness. This RCT on focal therapy versus usual care is urgently needed to enable focal therapy to overgrow the experimental status, provide the evidence needed for guidelines, and make this available for selected patients who benefit from this strategy. Because of its promising results in other countries, focal therapy is increasingly requested by patients, but due to the lack of high-quality evidence, it is not reimbursed yet. This has been designated by both the PCa patient support group and physicians as a failure of both the market and the funding agencies. The investigators, therefore, aim to perform a high-quality multi-center RCT to provide the evidence needed to decide on reimbursement and implementation of focal therapy in patients with intermediate-risk, unilateral clinically localized PCa in the Netherlands.

DETAILED DESCRIPTION:
In the Netherlands, most men with PCa are treated with radical whole-gland treatment, i.e. prostatectomy or a form of radiotherapy. The burden of complications such as incontinence and erectile dysfunction associated with radical treatment is considerable.

A recent systematic review by our group has shown that focal therapy of PCa seems to reduce the burden of treatment side-effects in men with intermediate-risk disease, maintaining their quality of life without compromising oncological effectiveness. The costs of side-effects that can be prevented are estimated at €5456 per patient, resulting in total expected cost savings of about €22 million per year in The Netherlands. Furthermore, exploration of the benefit-risk balance under patients showed that they are willing to sacrifice some survival for an improvement in quality of life (QoL).

Focal therapy comprises a modern alternative to selectively treat a specific part of the prostate while preserving the rest of the gland. There is, however, a lack of high-quality evidence, and numerous papers therefore recommend to perform a multicenter randomized controlled trial (RCT). The RCT should have long-term follow-up, predefined assessment of cancer-specific and health-related QoL outcome measures, and economic evaluations to inform policymakers regarding cost-effectiveness. This RCT on focal therapy versus usual care is urgently needed to enable focal therapy to overgrow the experimental status, provide the evidence needed for guidelines, and make this available for selected patients who benefit from this strategy. Because of its promising results in other countries, focal therapy is increasingly requested by patients, but due to the lack of high-quality evidence, it is not reimbursed yet. This has been designated by both the PCa patient support group and physicians as a failure of both the market and the funding agencies.

At present, all devices that are used in the proposed study are CE approved and no safety issues were reported in IDEAL stage 1 and 2a studies. For high-risk PCa, local radical therapy has been found to significantly improve oncological endpoints. However, for low- and intermediate-risk localized PCa, the different recommended options by guidelines (radical prostatectomy (RP), radiotherapy (RT), or active surveillance (AS)) have similar short- to medium-term oncological outcomes in randomized studies. A PROZIB database search and a KWF report showed that about 65% of the intermediate-risk patients that are eligible for focal therapy currently undergo either RP or RT. Furthermore, brachytherapy is only used to a limited extent (7%) in intermediate-risk patients in the Netherlands, and since it is not offered as a treatment option in the participating hospitals in this proposal, the investigators do not include this option in our study.

Active surveillance is mainly used for low-risk patients rather than for the intermediate-risk patients the investigators are aiming for in this study. Our systematic review concluded that more high-quality evidence is required before focal therapy can become available as a standard treatment. The majority of focal therapy studies were prospective development IDEAL stage 2a studies (feasibility studies), showing the limited adverse impact on functional outcomes and favorable oncological outcomes. Overall, focal therapy studies reported a median of 95% pad-free at 1-year and 85% of the patients had no clinically significant cancer in the treated area, respectively. High-quality multi-center comparative clinical trials, however, appear to be lacking. The appropriate management of patients with recurrent PCa following focal therapy has been an ongoing point of discussion. Marra et al. showed that evidence from assessments of salvage treatments after focal therapy failure is low and is derived from four retrospective salvage series. Available salvage options after focal therapy include RP and RT. Overall oncological outcomes are acceptable, although biochemical recurrence is slightly higher compared to primary PCa treatment, probably because of the higher aggressiveness of recurrent/persistent PCa. Functional outcomes and complications are not markedly worse compared to primary treatment. Salvage RP and salvage RT, therefore, seem feasible treatment options with acceptable oncological control and functional outcomes. Thus, re-treatment with salvage radiotherapy or salvage surgery remains a clinical option after focal therapy failure. Experience from other countries and our qualitative research on this topic taught us that many patients will consciously opt for an initial focal therapy to maintain their quality of life and because they can be treated later when deemed necessary with the other options.

All patients included in our trial will undergo intensive follow-up. Patients undergoing focal therapy will undergo quarterly PSA measurement and yearly prostate MRI, followed by a prostate biopsy after 12 months and thereafter if indicated based on the MRI. Since focal therapy is a one-time intervention, there will be no patients left in treatment or that require alternative fallback treatments. Ablation devices can be returned after the completion of the trial. The disposables are single-use and are depreciated. There are no specific costs associated with the discontinuation of focal treatment after the trial.

The investigators, therefore, aim to perform a high-quality multi-center RCT to provide the evidence needed to decide on reimbursement and implementation of focal therapy in patients with intermediate-risk, unilateral clinically localized PCa in the Netherlands. This study is funded by a national grant (Veelbelovende Zorg) from the Dutch Health Institute (Zorginstituut Nederland).

ELIGIBILITY:
Inclusion Criteria:

* Gleason score of 7 (3 + 4 or 4 + 3; ISUP grade 2/3)
* PSA level of ≤ 20 ng/ml
* Clinical stage ≤ T2b disease
* Life expectancy of ≥ 10 years
* Men with a prostate size ≤ 5 cm in sagittal length and ≤ 6 cm in axial length
* Fit, eligible, and normally destined for radical surgery or radiotherapy
* No concomitant cancer
* No previous treatment of their prostate
* An understanding of the Dutch language sufficient to receive written and verbal information about the trial, its consent process and the study questionnaires

Exclusion Criteria:

* Unfit for general anesthesia or radical surgery
* Low volume low-risk disease (≤4mm Gleason score of ≤ 6 / ISUP grade 1)
* High-risk disease (Gleason score of ≥ 8 / ISUP grade >3)
* Clinical T3 disease (extracapsular PCa)
* Men who have received previous active therapy for PCa.
* Men with evidence of extraprostatic disease.
* Men with an inability to tolerate a transrectal ultrasound.
* Cardiac pacemaker
* Metal implants/stents in the urethra or prostate.
* ASA ≥4
* Prostatic calcification/cysts that interfere with effective delivery of TULSA/HIFU based on MRCT.
* Men with renal impairment and a glomerular filtration rate (GFR) of < 30 ml/minute/1.73 m2.
* Unable to give consent to participate in the trial, as judged by the attending clinicians

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Oncological effectiveness (non-inferiority) defined as treatment failure | 36 months
  i.e. pathologically proven recurrent disease and/or the indication for retreatment with salvage treatment (RP, RT or systemic treatment or RT) in the focal therapy group and as biochemical recurrence and/or salvage treatment in the usual care group
Quality of life (superiority) measured with Functional Assessment of Cancer Therapy-Prostate questionnaire | 12 months
  Compare quality of life between the two arms measured with the FACT-P questionnaire. FACT-P scores of the subscales vary between 0-24 and 0-28, the total score is between 0-156. The higher the score, the better.

SECONDARY OUTCOMES:
Metastasis-free survival | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Metastasis-free survival as a validated surrogate endpoint of overall survival, comparing the proportion of patients between the arms who are free from metastatic disease.
Health-related quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for prostate cancer | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Compare quality of life measurements between the two arms using the EORTC QLQ-PR25 for sexual symptoms a higher score on the functional scales means a higher level of functioning, but on the symptomatic scales, a higher score means a greater severity of symptoms
Health-related quality of life using the International Consultation on Incontinence Questionnaire | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Quality of life measurements using the ICIQ-SF. Score ranges between1 and 21, a higher score means a greater severity of symptoms.
Health-related quality of life regarding urinary symptoms using the International Prostate Symptom Score questionnaire | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Compare quality of life measurements between the two arms using the IPSS The score ranges between 0 and 35, a higher score means a greater severity of symptoms
Health-related quality of life using the Sexual Health Inventory for Men International Index of Erectile Function-5 questionnaire | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Compare quality of life measurements between the two arms regarding sexual function using the SHIM IIEF-5 questionnaire, the score ranges between 8 and 25, a higher score means lesser severity of symptoms.
Health-related quality of life using the 5-dimension health-related quality of life from the uroQol group | at baseline, 3, 6, 12, 24, 36, 48 and 60 months
  Quality of life measurements regarding mobility, self-care, usual activities, pain/discomfort, anxiety/depression using the EuroQol 5D 5level questionnaire
Disease progression | 60 months
Disease specific mortality | 60 months
  Compare the mortality between the two arms regarding prostate cancer
All-cause mortality | 60 months
  Compare the overall mortality between the two arms.
Operating time | Immediately after the procedure
  Compare the total time of the procedure between the two arms.
Hospital care stay | Immediately after procedure
  Compare the length of the hospital stay between the two arms.
Pathology results after biopsy and/or radical prostatectomy | 60 months
  • Pathology results after biopsy and/or radical prostatectomy will be summarized using descriptive statistics, primarily the frequency and proportion of events.
Adverse events | 60 months
  • Treatment-related complications will be recorded according to the Clavien-Dindo classification. We will calculate both an overall mean risk difference and 95% confidence interval as well as a mean risk difference per item, and their corresponding 95% CI
Cost-effectiveness will be measured using the iMTA Medical Consumption Questionnaire | 60 months
  Costs will be calculated according to the Dutch guideline for costing research, by multiplying resource use with the corresponding unit costs. Average costs will be calculated in both groups, and differences will be calculated inclusive of 95% confidence intervals. Effectiveness will be measured in terms of quality-adjusted life years (QALYs).
Cost-effectiveness will be measured using the IMTA Productivity Cost Questionnaire | 60 months
  Costs will be calculated according to the Dutch guideline for costing research, by multiplying resource use with the corresponding unit costs. Average costs will be calculated in both groups, and differences will be calculated inclusive of 95% confidence intervals. Effectiveness will be measured in terms of quality-adjusted life years (QALYs).

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - Radboud University Medical Centre, Nijmegen, Gelderland
  - Hifu kliniek, Etten-Leur, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - Isala klinieken, Zwolle, Overijssel
  - St. Antonius hospital, Nieuwegein, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haglind E, Carlsson S, Stranne J, Wallerstedt A, Wilderang U, Thorsteinsdottir T, Lagerkvist M, Damber JE, Bjartell A, Hugosson J, Wiklund P, Steineck G; LAPPRO steering committee. Urinary Incontinence and Erectile Dysfunction After Robotic Versus Open Radical Prostatectomy: A Prospective, Controlled, Nonrandomised Trial. Eur Urol. 2015 Aug;68(2):216-25. doi: 10.1016/j.eururo.2015.02.029. Epub 2015 Mar 12. PMID 25770484
- [Background] Hopstaken JS, Bomers JGR, Sedelaar MJP, Valerio M, Futterer JJ, Rovers MM. An Updated Systematic Review on Focal Therapy in Localized Prostate Cancer: What Has Changed over the Past 5 Years? Eur Urol. 2022 Jan;81(1):5-33. doi: 10.1016/j.eururo.2021.08.005. Epub 2021 Sep 4. PMID 34489140
- [Background] de Bekker-Grob EW, Bliemer MC, Donkers B, Essink-Bot ML, Korfage IJ, Roobol MJ, Bangma CH, Steyerberg EW. Patients' and urologists' preferences for prostate cancer treatment: a discrete choice experiment. Br J Cancer. 2013 Aug 6;109(3):633-40. doi: 10.1038/bjc.2013.370. Epub 2013 Jul 16. PMID 23860533
- [Background] Watson V, McCartan N, Krucien N, Abu V, Ikenwilo D, Emberton M, Ahmed HU. Evaluating the Trade-Offs Men with Localized Prostate Cancer Make between the Risks and Benefits of Treatments: The COMPARE Study. J Urol. 2020 Aug;204(2):273-280. doi: 10.1097/JU.0000000000000754. Epub 2020 Jan 22. PMID 31967521
- [Background] Blazevski A, Scheltema MJ, Yuen B, Masand N, Nguyen TV, Delprado W, Shnier R, Haynes AM, Cusick T, Thompson J, Stricker P. Oncological and Quality-of-life Outcomes Following Focal Irreversible Electroporation as Primary Treatment for Localised Prostate Cancer: A Biopsy-monitored Prospective Cohort. Eur Urol Oncol. 2020 Jun;3(3):283-290. doi: 10.1016/j.euo.2019.04.008. Epub 2019 May 16. PMID 31103721
- [Background] Chin JL, Billia M, Relle J, Roethke MC, Popeneciu IV, Kuru TH, Hatiboglu G, Mueller-Wolf MB, Motsch J, Romagnoli C, Kassam Z, Harle CC, Hafron J, Nandalur KR, Chronik BA, Burtnyk M, Schlemmer HP, Pahernik S. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue in Patients with Localized Prostate Cancer: A Prospective Phase 1 Clinical Trial. Eur Urol. 2016 Sep;70(3):447-55. doi: 10.1016/j.eururo.2015.12.029. Epub 2016 Jan 6. PMID 26777228
- [Background] Bonekamp D, Wolf MB, Roethke MC, Pahernik S, Hadaschik BA, Hatiboglu G, Kuru TH, Popeneciu IV, Chin JL, Billia M, Relle J, Hafron J, Nandalur KR, Staruch RM, Burtnyk M, Hohenfellner M, Schlemmer HP. Twelve-month prostate volume reduction after MRI-guided transurethral ultrasound ablation of the prostate. Eur Radiol. 2019 Jan;29(1):299-308. doi: 10.1007/s00330-018-5584-y. Epub 2018 Jun 25. PMID 29943185
- [Background] Ramsay E, Mougenot C, Staruch R, Boyes A, Kazem M, Bronskill M, Foster H, Sugar L, Haider M, Klotz L, Chopra R. Evaluation of Focal Ablation of Magnetic Resonance Imaging Defined Prostate Cancer Using Magnetic Resonance Imaging Controlled Transurethral Ultrasound Therapy with Prostatectomy as the Reference Standard. J Urol. 2017 Jan;197(1):255-261. doi: 10.1016/j.juro.2016.06.100. Epub 2016 Aug 18. PMID 27545572
- [Background] Marra G, Valerio M, Emberton M, Heidenreich A, Crook JM, Bossi A, Pisters LL. Salvage Local Treatments After Focal Therapy for Prostate Cancer. Eur Urol Oncol. 2019 Sep;2(5):526-538. doi: 10.1016/j.euo.2019.03.008. Epub 2019 Apr 15. PMID 31412013
- [Background] Nathan A, Ng A, Mitra A, Sooriakumaran P, Davda R, Patel S, Fricker M, Kelly J, Shaw G, Rajan P, Sridhar A, Nathan S, Payne H. Comparative Effectiveness Analyses of Salvage Prostatectomy and Salvage Radiotherapy Outcomes Following Focal or Whole-Gland Ablative Therapy (High-Intensity Focused Ultrasound, Cryotherapy or Electroporation) for Localised Prostate Cancer. Clin Oncol (R Coll Radiol). 2022 Jan;34(1):e69-e78. doi: 10.1016/j.clon.2021.10.012. Epub 2021 Nov 3. PMID 34740477
- [Background] Gharzai LA, Jiang R, Wallington D, Jones G, Birer S, Jairath N, Jaworski EM, McFarlane MR, Mahal BA, Nguyen PL, Sandler H, Morgan TM, Reichert ZR, Alumkal JJ, Mehra R, Kishan AU, Fizazi K, Halabi S, Schaeffer EM, Feng FY, Elliott D, Dess RT, Jackson WC, Schipper MJ, Spratt DE. Intermediate clinical endpoints for surrogacy in localised prostate cancer: an aggregate meta-analysis. Lancet Oncol. 2021 Mar;22(3):402-410. doi: 10.1016/S1470-2045(20)30730-0. PMID 33662287
- [Background] Skolarus TA, Dunn RL, Sanda MG, Chang P, Greenfield TK, Litwin MS, Wei JT; PROSTQA Consortium. Minimally important difference for the Expanded Prostate Cancer Index Composite Short Form. Urology. 2015 Jan;85(1):101-5. doi: 10.1016/j.urology.2014.08.044. PMID 25530370
- [Background] Tay KJ, Scheltema MJ, Ahmed HU, Barret E, Coleman JA, Dominguez-Escrig J, Ghai S, Huang J, Jones JS, Klotz LH, Robertson CN, Sanchez-Salas R, Scionti S, Sivaraman A, de la Rosette J, Polascik TJ. Patient selection for prostate focal therapy in the era of active surveillance: an International Delphi Consensus Project. Prostate Cancer Prostatic Dis. 2017 Sep;20(3):294-299. doi: 10.1038/pcan.2017.8. Epub 2017 Mar 28. PMID 28349978
- [Background] Cella D, Nichol MB, Eton D, Nelson JB, Mulani P. Estimating clinically meaningful changes for the Functional Assessment of Cancer Therapy--Prostate: results from a clinical trial of patients with metastatic hormone-refractory prostate cancer. Value Health. 2009 Jan-Feb;12(1):124-9. doi: 10.1111/j.1524-4733.2008.00409.x. Epub 2008 Jul 18. PMID 18647260